CLINICAL TRIAL: NCT03312127
Title: Evaluation of Peri-surgical Results at Short and Mean Terms of the GORE ® Excluder Iliac Branch Endoprosthesis
Acronym: HYPOGRAFT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: End of inclusion period
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14 7427 15
Record Dates: First submitted 2017-07-27; First posted 2017-10-17 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Iliac Aneurysm
MeSH Terms: conditions — Iliac Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GORE Excluder (Experimental): GORE Excluder Iliac Branch Endoprosthesis arm with 'ILIAC ENDOPROSTHESIS GORE EXCLUDER'
  Interventions: Device: ILIAC ENDOPROSTHESIS GORE EXCLUDER

INTERVENTIONS:
Device: ILIAC ENDOPROSTHESIS GORE EXCLUDER — Set up of GORE ® Excluder Iliac Branch Endoprosthesis in endovascular barring of complex aneurysms without distal neck. In the immediate post-operating follow-up visit and at the 3 months visit and the 12 months visit after surgery, an ultra-sound scan, a tomodensitometric exam and a walking test on a treadmill with oximetric gluteal region exploration will systematically be performed.

SUMMARY:
The aim of this project is to demonstrate the benefit of the use of aortic iliac branch endoprosthesis in the iliac aneurysms and to avoid the classic complications.

ELIGIBILITY:
Inclusion Criteria:

* High surgical risk:

  * Comorbidity cardiopulmonary
  * Renal insufficiency
  * Hostile abdomen including ascites or portal hypertension
* Anatomic criteria:

  * Primitive iliac aneurysm superior to 25 mm without collar
  * Primitive iliac length superior to 40 mm
  * Primitive iliac distal diameter superior to 14 mm
  * Presence of internal iliac collar
* Affiliation to a social security system

Exclusion Criteria:

* Patient without surgical risk
* Non-respect of the Anatomic criteria
* Patient with known allergy to the materials of the device
* Patient with systemic infection
* Patient with severe renal insufficiency
* Patient unable to complete the oximetry test
* Persons under legal protection

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-07-26 (Actual); Study Completion 2018-07-26 (Actual)

PRIMARY OUTCOMES:
Primary permeability maintenance of the iliac branch endoprosthesis, following its insertion (binary criterion) | At the immediate post-operating follow-up visit
  Primary permeability maintenance of the iliac branch endoprosthesis, following its insertion. It is a binary criterion (permeable or not) This criterion will be evaluated by a doppler ultrasound. These exams will be performed by a unique vascular physician, who will measure the hemodynamic criterions and the associated gluteal region oximetry.
  Endoprosthesis will be considered to be permeable if the patient is asymptomatic (absence of gluteal claudication), if Doppler ultrasound and angio-scan confirm the permeability of the endoprosthesis.
Primary permeability maintenance of the iliac branch endoprosthesis, following its insertion (binary criterion) | at 3 months after surgery
  Primary permeability maintenance of the iliac branch endoprosthesis, following its insertion. It is a binary criterion (permeable or not) This criterion will be evaluated by a doppler ultrasound. These exams will be performed by a unique vascular physician, who will measure the hemodynamic criterions and the associated gluteal region oximetry.
  Endoprosthesis will be considered to be permeable if the patient is asymptomatic (absence of gluteal claudication), if Doppler ultrasound and angio-scan confirm the permeability of the endoprosthesis.
Primary permeability maintenance of the iliac branch endoprosthesis, following its insertion (binary criterion) | at 12 months after surgery
  Primary permeability maintenance of the iliac branch endoprosthesis, following its insertion. It is a binary criterion (permeable or not) This criterion will be evaluated by a doppler ultrasound. These exams will be performed by a unique vascular physician, who will measure the hemodynamic criterions and the associated gluteal region oximetry.
  Endoprosthesis will be considered to be permeable if the patient is asymptomatic (absence of gluteal claudication), if Doppler ultrasound and angio-scan confirm the permeability of the endoprosthesis.
  Primary permeability will be considered non-maintained at 1 year if a stenosis >70% or a thrombosis of the hypogastric branch is observed by ultra-sound scan at a follow-up visit during the first year after surgery or at a ultra-sound scan exam motivated by pelvic ischemia clinical signs

SECONDARY OUTCOMES:
Morbidity | peri-operative, at short term (3 months), mean-term (12 months)
  Evaluation of the morbidity:
  * Minor events (no revision surgery needed):
    * General: pulmonary, cardiologic, renal
    * Local: hematoma, false aneurysm, Impaired wound healing
  * Major events (revision surgery needed):
    * Endoleak
    * Thrombosis
    * Rupture

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre BOSSAVY, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: Undecided